CLINICAL TRIAL: NCT03366935
Title: Combined Implementation of Dural Puncture Epidural Technique and Programmed Intermittent Epidural Bolus for Labor Analgesia
Brief Title: Combined Implementation of Dural Puncture Epidural and Programmed Intermittent Epidural Bolus for Labor Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: anesthesia dapartment
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Labor Pain; Labor Analgesia
Keywords: labor analgesia; dural puncture epidural (DPE); standard Epidural (EPL); continuous epidural infusion (CEI); programmed intermittent epidural bolus (PIEB)
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EPL and CEI (Experimental): Those with receive a standard epidural (EPL) and continuous epidural infusion(CEI) + patient-controlled epidural analgesia (PCEA)
  Interventions: Other: EPL and CEI
- DPE and CEI (Active Comparator): Those with receive a dural puncture labor epidural (DPE) and continuous epidural infusion(CEI) + patient-controlled epidural analgesia (PCEA)
  Interventions: Other: DPE and CEI
- DPE and PIEB (Active Comparator): Those with receive a dural puncture labor epidural (DPE) and programmed intermittent epidural boluses(PIEB) + patient-controlled epidural analgesia (PCEA)
  Interventions: Other: DPE and PIEB

INTERVENTIONS:
Other: EPL and CEI — Procedure: Standard epidural placement(EPL)
  Drug: ropivacaine Drug: sufentani 0.1% ropivacaine + sufentanil 0.3μg/mL
  Device: Infusion pump Infusion pump set to continuous epidural infusion(CEI) plus patient-controlled epidural analgesia (PCEA).
  Arms: EPL and CEI
Other: DPE and CEI — Procedure: Dural puncture epidural (DPE) Epidural with spinal needle placed to create a single dural puncture and confirm free flow of cerebral spinal fluid (CSF) , without direct medication administration into the subarachnoid space.
  Drug: ropivacaine Drug: sufentani 0.1% ropivacaine + sufentanil 0.3μg/mL
  Device: Infusion pump Infusion pump set to continuous epidural infusion(CEI) plus patient-controlled epidural analgesia (PCEA).
  Arms: DPE and CEI
Other: DPE and PIEB — Procedure: Dural puncture epidural (DPE) Epidural with spinal needle placed to create a single dural puncture and confirm free flow of cerebral spinal fluid (CSF) , without direct medication administration into the subarachnoid space.
  Drug: ropivacaine Drug: sufentani 0.1% ropivacaine + sufentanil 0.3μg/mL
  Device: Infusion pump Infusion pump set to programmed intermittent epidural boluses (PIEB) plus patient-controlled epidural analgesia (PCEA).
  Arms: DPE and PIEB

SUMMARY:
This study intends to carry out a prospective, randomized double-blind study to evaluate the safety and efficacy of the combined implementation of Dural puncture epidural (DPE) technique and Programmed intermittent epidural bolus (PIEB) for labor analgesia.

DETAILED DESCRIPTION:
Epidural (EPL) technique is the standard technique for labor analgesia, but can be associated with slow onset and inadequate sacral spread, unilateral or patchy sensory blockade, motor impairment. The combined spinal epidural (CSE) technique can provide rapid onset of analgesia, but is associated with greater side effects, including pruritus, fetal bradycardia and delayed testing of epidural catheters. Dural puncture epidural (DPE) technique is a modification of CSE technique. A spinal needle is introduced through the epidural needle to create a single dural puncture , after intrathecal space was identified by the free flow of cerebrospinal fluid (CSF) , the needle was removed without direct medication administration into the subarachnoid space. Privous studies have demonstrated that the DPE technique can improve block quality over the EPL technique with fewer maternal and fetal side effects than the CSE technique for parturients requesting labor analgesia. Besides the neuraxial techniques, maintenance regimens is another factor that affect the analgesic effect. Programmed intermittent epidural bolus (PIEB) provides greater spread of local anesthetic solution within the epidural space and therefore superior quality of analgesia compared with continuous epidural infusion (CEI). We designed this prospective randomized, double-blind study to evaluate the safety and efficacy of the combined implementation of DPE technique and PIEB for labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. women requeste labor analgesia
2. ASA I or II
3. at 37-42 weeks' gestation
4. nulliparous
5. singleton pregnancy, vertex presentation
6. visual Numerical Rating Scale (VNRS) at requesting analgesia > 5 (NRPS 0-10)
7. cervical dilatation < 5 cm

Exclusion Criteria:

1. patient refusal to participate in the study
2. age <20 years or >40 years
3. body mass Index(BMI)>50 (Kg/m2)
4. clinically significant diseases of pregnancy (i.e.,gestational hypertension, preeclampsia, gestational placenta previa, placental abruption diabetes)
5. contraindications to neuraxial analgesia
6. drug abuse
7. conditions associated with an increased risk of a cesarean delivery (i.e., history of uterine anomaly or surgery, morbid obesity) and known anomalies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant patients
Enrollment: 120 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Compare time of onset of labor analgesia among the study groups | From epidural infusion initiate to delivery
  Visual Numerical Rating Scale (VNRS) ≤ 10 mm on a 100-mm scale

SECONDARY OUTCOMES:
Incidence of side effect | 24 hours post delivery
  maternal hypotension,fetal bradycardia, maternal motor block,post-dural puncture headache,nausea, vomiting,pruritus,nerve damage
Sensory block level | 24 hours post delivery
  Sensory block will be assessed bilaterally
Total anesthetic dose required | From epidural infusion initiate to 1h post delivery
  Including physician interventions, programmed doses, and patient controlled doses
Mode of delivery | From epidural infusion initiate to delivery
  Spontaneous, Instrumental, or cesarean delivery
Apgar scores | 30 mins post delivery
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are skin color, pulse rate, reflex irritability grimace, activity and respiratoty effort

CONTACTS AND LOCATIONS:
Overall Officials: YuJie Song, MD, Study Chair — Department of Anesthesiaology, Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai First Maternity and Infant Hospital, Tongji University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norris MC, Fogel ST, Conway-Long C. Combined spinal-epidural versus epidural labor analgesia. Anesthesiology. 2001 Oct;95(4):913-20. doi: 10.1097/00000542-200110000-00020. PMID 11605932
- [Background] Eappen S, Blinn A, Segal S. Incidence of epidural catheter replacement in parturients: a retrospective chart review. Int J Obstet Anesth. 1998 Oct;7(4):220-5. doi: 10.1016/s0959-289x(98)80042-3. PMID 15321183
- [Background] Groden J, Gonzalez-Fiol A, Aaronson J, Sachs A, Smiley R. Catheter failure rates and time course with epidural versus combined spinal-epidural analgesia in labor. Int J Obstet Anesth. 2016 May;26:4-7. doi: 10.1016/j.ijoa.2016.01.004. Epub 2016 Jan 14. PMID 26971650
- [Background] Suzuki N, Koganemaru M, Onizuka S, Takasaki M. Dural puncture with a 26-gauge spinal needle affects spread of epidural anesthesia. Anesth Analg. 1996 May;82(5):1040-2. doi: 10.1097/00000539-199605000-00028. PMID 8610864
- [Background] Cappiello E, O'Rourke N, Segal S, Tsen LC. A randomized trial of dural puncture epidural technique compared with the standard epidural technique for labor analgesia. Anesth Analg. 2008 Nov;107(5):1646-51. doi: 10.1213/ane.0b013e318184ec14. PMID 18931227
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Background] Wilson SH, Wolf BJ, Bingham K, Scotland QS, Fox JM, Woltz EM, Hebbar L. Labor Analgesia Onset With Dural Puncture Epidural Versus Traditional Epidural Using a 26-Gauge Whitacre Needle and 0.125% Bupivacaine Bolus: A Randomized Clinical Trial. Anesth Analg. 2018 Feb;126(2):545-551. doi: 10.1213/ANE.0000000000002129. PMID 28622178
- [Background] Patkar CS, Vora K, Patel H, Shah V, Modi MP, Parikh G. A comparison of continuous infusion and intermittent bolus administration of 0.1% ropivacaine with 0.0002% fentanyl for epidural labor analgesia. J Anaesthesiol Clin Pharmacol. 2015 Apr-Jun;31(2):234-8. doi: 10.4103/0970-9185.155155. PMID 25948908
- [Background] McKenzie CP, Cobb B, Riley ET, Carvalho B. Programmed intermittent epidural boluses for maintenance of labor analgesia: an impact study. Int J Obstet Anesth. 2016 May;26:32-8. doi: 10.1016/j.ijoa.2015.11.005. Epub 2015 Nov 27. PMID 26775896
- [Background] Carvalho B, George RB, Cobb B, McKenzie C, Riley ET. Implementation of Programmed Intermittent Epidural Bolus for the Maintenance of Labor Analgesia. Anesth Analg. 2016 Oct;123(4):965-71. doi: 10.1213/ANE.0000000000001407. PMID 27464978
- [Background] Fettes PD, Moore CS, Whiteside JB, McLeod GA, Wildsmith JA. Intermittent vs continuous administration of epidural ropivacaine with fentanyl for analgesia during labour. Br J Anaesth. 2006 Sep;97(3):359-64. doi: 10.1093/bja/ael157. Epub 2006 Jul 18. PMID 16849382
- [Derived] Song Y, Du W, Zhou S, Zhou Y, Yu Y, Xu Z, Liu Z. Effect of Dural Puncture Epidural Technique Combined With Programmed Intermittent Epidural Bolus on Labor Analgesia Onset and Maintenance: A Randomized Controlled Trial. Anesth Analg. 2021 Apr 1;132(4):971-978. doi: 10.1213/ANE.0000000000004768. PMID 32282386